CLINICAL TRIAL: NCT02691338
Title: Monitoring Neurological Deterioration in Anaesthetised Patients With Electroencephalogram (EEG): Demonstration With Patients Undergoing Neurovascular Intervention After Cerebrovascular Attack (CVA).
Brief Title: Monitoring Neurological Deterioration in Anaesthetised Patients With Electroencephalogram (EEG)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0459-15-Rambam-CTIL
Record Dates: First submitted 2016-02-09; First posted 2016-02-25 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: CVA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients undergoing thrombectomy: 150 anesthetized patients undergoing intra-arterial catheterization for thrombectomy after CVA. The patients will be recruited at the Rambam Health Center, Haifa, Israel. The patients will undergo EEG recording during the procedure, without changing patient's standard treatment care. The EEG recording will continue after the procedure for four hours approximately, while the patients are admitted to intensive care unit (ICU).
  Interventions: Other: EEG; Other: Routine follow up tests
- Control - healthy individuals: 20 health individuals under general anesthesia or sedation for other surgery or procedures. They will undergo EEG recording during the surgery/ procedure, to validate the sensitivity of the EEG to the effect of the anaesthetic medications.
  Interventions: Other: EEG

INTERVENTIONS:
Other: EEG — EEG analysis
Other: Routine follow up tests — Routine tests for patients after CVA. This include: neurologic evaluation, Brain CT, Angiography
  Groups: patients undergoing thrombectomy

SUMMARY:
The incidence of perioperative stroke in the non-cardiac, non-vascular, non-neurological high risk surgical population is 2%. It is higher (~5%) for cardiac surgery and carotid endarterectomy patients, with a stroke associated mortality of up to 60%. These patients could be immediately treated if their condition was detected on time. Currently, there is no standard brain monitoring procedure for anaesthetised patients. The purpose of the proposed study is to optimize and validate an online monitor for neurological deterioration under anaesthesia based on an easily operatable EEG system comprised of 4 electrodes, a reference electrode and a newely developed algorithm for analyzing the EEG signal. The monitor aims at generating an immediate warning at the onset of neurological deterioration. For the purpose of technology development with a minimal sample size, it is necessary to select a patient population that demonstrates significant neurological dynamics under anaesthesia. We will therefore focus on anesthesized patients undergoing neurovascular thrombectomy after CVA.

DETAILED DESCRIPTION:
The research aim is to validate a novel ground-breaking and easy-to-use EEG-based algorithm for sensing cerebrovascular accident (CVA) events under anaesthesia. Today there is no standard tool for CVA detection in anaesthetized patients. Thus the possibility of waking up from anaesthesia with severe brain damage is devastating. Patients undergoing cardiac surgery (such as valve replacement, CABG, thoracic aorta replacement, PTCA, TAVI (trans-aortic valve implantation)), carotid endarterectomy and surgery in sitting position, are at exceptionally high risk. We have developed a unique algorithm for detecting brain ischemia in anaesthetized patients, based on data acquired from 4 EEG electrodes. Our final goal is to develop a system that triggers an alarm when an ischemia occurs in an anaesthetized patient and during the peri-operative period.

In order to validate and optimize our system, we require a small sample size to test and validate the technology. The population for this study includes patients with acute CVA who undergo mechanical thrombectomy under anaesthesia. Although these patients already have CVA, clinical dynamics is high in this population, and will enable a demonstration of our ability to recognize immediate changes in neurological status (improvement or deterioration).

We believe this innovative EEG based system could be of major significance to millions of patients annually.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent (by individual or guardian)
* Undergoing thrombectomy procedure under anaesthesia for acute CVA
* for control:
* Healthy individual, with no neurological disease undergoing sedation for procedure

Exclusion Criteria:

* Age < 18 years
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CVA undergoing percutaneous thrombectomy under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-02; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
EEG-based interhemispheric synchronization index | Interhemispheric synchronization is measured retrospectively - for the whole period the patient is under general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Dana Baron Shahaf, MD PhD, Study Director — Rambam Health Care Center
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahaf DB, Shahaf G, Mehta J, Venkatraghavan L. Intracarotid Etomidate Decreases the Interhemispheric Synchronization in Electroencephalogram (EEG) During the Wada Test. J Neurosurg Anesthesiol. 2016 Oct;28(4):341-6. doi: 10.1097/ANA.0000000000000241. PMID 26536542
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Moritz S, Kasprzak P, Arlt M, Taeger K, Metz C. Accuracy of cerebral monitoring in detecting cerebral ischemia during carotid endarterectomy: a comparison of transcranial Doppler sonography, near-infrared spectroscopy, stump pressure, and somatosensory evoked potentials. Anesthesiology. 2007 Oct;107(4):563-9. doi: 10.1097/01.anes.0000281894.69422.ff. PMID 17893451
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Background] Foreman B, Claassen J. Quantitative EEG for the detection of brain ischemia. Crit Care. 2012 Dec 12;16(2):216. doi: 10.1186/cc11230. No abstract available. PMID 22429809
- [Background] Shahaf G, Pratt H. Thorough specification of the neurophysiologic processes underlying behavior and of their manifestation in EEG - demonstration with the go/no-go task. Front Hum Neurosci. 2013 Jun 24;7:305. doi: 10.3389/fnhum.2013.00305. eCollection 2013. PMID 23805094
- [Background] Shahaf G, Fisher T, Aharon-Peretz J, Pratt H. Comprehensive analysis suggests simple processes underlying EEG/ERP - demonstration with the go/no-go paradigm in ADHD. J Neurosci Methods. 2015 Jan 15;239:183-93. doi: 10.1016/j.jneumeth.2014.10.016. Epub 2014 Nov 1. PMID 25445244